CLINICAL TRIAL: NCT00891228
Title: A Multicenter, Randomized, Double-Blind Comparator Trial of the Safety and Sperm and Gonadotropin Suppression Resulting From Combined Use of Nestorone® Gel (0, 8 or 12 mg NES) and Testosterone Gel (10 g) Compared With Testosterone Gel in Normal Men
Brief Title: Study of the Safety, and Sperm and Gonadotropin Suppression of a Contraceptive Gel in Normal Men
Acronym: CCN007
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Premier Research (Other)
Collaborators: Population Council (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CCN007
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Results first posted 2018-05-24 (Actual); Last update posted 2018-05-24 (Actual); Status verified 2018-04

CONDITIONS: Contraception
Keywords: Contraception; Male Contraception; Suppression of Sperm Production
MeSH Terms: interventions — Testosterone; ST 1435

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Testosterone Gel 10 g and Nestorone® 0 mg per day (Placebo Comparator): Two individual packets of Testosterone Gel, each with 5 g of gel applied to each arm delivering a total of 100 mg of Testosterone on the skin. Nestorone® Gel will be delivered by a pump configured to deliver 4 mL of gel containing 0 mg of Nestorone® by pressing two times with the 2 mL dispenser head.
  Interventions: Drug: Testosterone; Drug: Nestorone®
- Testosterone Gel 10 g and Nestorone® 8 mg per day (Experimental): Two individual packets of Testosterone Gel, each with 5 g of gel applied to each arm delivering a total of 100 mg of Testosterone on the skin. Nestorone® Gel will be delivered by a pump configured to deliver a metered volume of Nestorone® Gel containing 8 mg of Nestorone®. For 8 mg Nestorone® dose; Nestorone® Gel will be delivered in 4 mL volume (2 mg NES mL gel) by pressing two times with 2 mL dispenser head.
  Interventions: Drug: Testosterone; Drug: Nestorone®
- Testosterone Gel 10 g plus Nestorone® Gel 12 mg per day (Experimental): Two individual packets of Testosterone Gel, each with 5 g of gel applied to each arm delivering a total of 100 mg of Testosterone on the skin. Nestorone® Gel will be delivered by a pump configured to deliver a metered volume of Nestorone® Gel containing 12 mg of Nestorone®. For 12 mg Nestorone® dose; Nestorone® Gel will be delivered in 4 mL volume (3 mg Nestorone®/mL gel) by pressing two times with 2 mL dispenser head.
  Interventions: Drug: Testosterone; Drug: Nestorone®

INTERVENTIONS:
Drug: Testosterone — Two individual packets of T Gel, each with 5 g of gel applied to each arm delivering a total of 100 mg of T on the skin daily.
Drug: Nestorone® — Nestorone® Gel will be delivered by a pump configured to deliver a metered volume of Nestorone® Gel containing 8 mg of Nestorone®. For 8 mg Nestorone® dose; Nestorone® Gel will be delivered in 4 mL volume (2 mg Nestorone® mL gel) by pressing two times with 2 mL dispenser head.
  Arms: Testosterone Gel 10 g and Nestorone® 8 mg per day
Drug: Nestorone® — Nestorone® Gel will be delivered by a pump configured to deliver a metered volume of Nestorone® Gel containing 12 mg of Nestorone®. For 12 mg Nestorone® dose; Nestorone® Gel will be delivered in 4 mL volume (3 mg Nestorone®/mL gel) by pressing two times with 2 mL dispenser head.
  Arms: Testosterone Gel 10 g plus Nestorone® Gel 12 mg per day
Drug: Nestorone® — Nestorone® Gel will be delivered by a pump configured to deliver 4 mL of gel containing 0 mg of Nestorone® by pressing two times with the 2 mL dispenser head.
  Arms: Testosterone Gel 10 g and Nestorone® 0 mg per day

SUMMARY:
To determine the number of men who have suppression of sperm production when using a daily regimen of Nestorone® Gel (0, 8 or 12 mg) and Testosterone Gel applied transdermally.

ELIGIBILITY:
Inclusion Criteria

Men who meet all the following criteria are eligible for enrollment in the trial:

1. Male volunteers in good health as confirmed by physical examination, medical history, and clinical laboratory tests of blood and urine at the time of screening
2. 18 to 50 years of age
3. BMI ≤ 33 calculated as weight in Kg/ (height in cm) 2
4. No history of hormonal therapy use in the last six months prior to the first screening visit
5. Subject will agree to use a recognized effective method of contraception with his partner (i.e. at a minimum, use double-barrier contraception) during the course of the study treatment and recovery phase
6. In the opinion of the investigator, subject is able to comply with the protocol, understand and sign an informed consent and HIPAA form
7. Does not meet any of the exclusion criteria.

Exclusion Criteria:

Men who meet any of the following criteria are NOT eligible for enrollment in the trial:

1. Men participating in another clinical trial involving an investigational drug within the last 30 days prior to the first screening visit
2. Men not living in the catchment's area of the clinic or within a reasonable distance from the site
3. Clinically significant abnormal findings at screening
4. Elevated PSA (levels ≥ 4 ng/mL), according to local laboratory normal values
5. Abnormal serum chemistry values, according to local laboratory normal values that indicate liver or kidney dysfunction or that may be considered clinically significant. Other abnormal lab values may also be exclusionary, at the discretion of the investigator
6. Sperm concentration below 15 million/mL in more than one of three screening samples
7. Use of androgens or body building substances within 6 months before first screening visit
8. Diastolic (D) blood pressure (BP) ≥ 85 and Systolic (S) BP ≥ 135 mm Hg; (BP will be taken 3 times at 5 minute intervals and the mean of all measurements be considered)
9. History of hypertension, including hypertension controlled with treatment
10. Known history of primary testicular disease or disorders of the hypothalamic-pituitary axis
11. Known hypersensitivity to progestins
12. Family or personal history of venous thromboembolism
13. Benign or malignant liver tumors; active liver disease
14. History of breast carcinoma
15. Known history of reproductive dysfunction including vasectomy or infertility
16. Known history of cardiac, renal, hepatic or prostatic disease
17. A serious systemic disease such as diabetes mellitus or morbid obesity (body weight greater than 120% of ideal body weight or BMI limitation as above)
18. History of sleep apnea
19. Known or suspected alcoholism or drug abuse that may affect metabolism/transformation of steroid hormones and study treatment compliance
20. Known dermatitis or severe skin disorder
21. Partner is known to be pregnant
22. Men desiring fertility within the first 24 weeks of study participation.

Men participating in competitive sports where drug screening for prohibited substances (including anabolic steroids) is routine will be advised of the relative and temporary hazards that participating in this study may have for their fertility or sporting status.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2009-05; Primary Completion 2010-05 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Wang, MD, Principal Investigator — LA BioMedical Research Institute, Harbor-UCLA; William Bremner, MD, PhD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Los Angeles Biomedical Research Institute at Harbor-UCLA, Torrance, California
  - University of Washington, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Testosterone Gel 10 g and Nestorone® 0 mg Per Day | Testosterone Gel 10 g and Nestorone® 8 mg Per Day | Testosterone Gel 10 g Plus Nestorone® Gel 12 mg Per Day
Started | 32 | 33 | 34
Completed | 21 | 20 | 19
Not Completed | 11 | 13 | 15
Not completed — Adverse Event | 0 | 2 | 3
Not completed — Withdrawal by Subject | 2 | 4 | 5
Not completed — Protocol Violation | 3 | 1 | 2
Not completed — Physician Decision | 2 | 1 | 0
Not completed — Lost to Follow-up | 4 | 4 | 5
Not completed — Pregnancy | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Testosterone Gel 10 g and Nestorone® 0 mg Per Day | Testosterone Gel 10 g and Nestorone® 8 mg Per Day | Testosterone Gel 10 g Plus Nestorone® Gel 12 mg Per Day | Total
Number analyzed (Participants) | 32 | 33 | 34 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 32 | 33 | 34 | 99
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 32 | 33 | 34 | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 9 | 10 | 27
  Not Hispanic or Latino | 24 | 24 | 24 | 72
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 7 | 1 | 1 | 9
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 0 | 3
  Black or African American | 5 | 3 | 7 | 15
  White | 16 | 24 | 25 | 65
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 32 | 33 | 34 | 99

OUTCOME MEASURES:

1. Primary Outcome: The Number of Men Who Have Suppression of Sperm Production ≤1Million/mL Million/mL When Using a Daily Regimen of Nestorone® Gel (0, 8 or 12 mg) and Testosterone Gel Applied Transdermally.
Time Frame: 24 Weeks
Measure: Number; unit: participants
Arm/Group | Testosterone Gel 10 g and Nestorone® 0 mg Per Day | Testosterone Gel 10 g and Nestorone® 8 mg Per Day | Testosterone Gel 10 g Plus Nestorone® Gel 12 mg Per Day
Number analyzed (Participants) | 22 | 18 | 16
participants | 5 | 15 | 13

2. Secondary Outcome: The Number of Men Who Have Suppression of Sperm Production ≤3 Million/mL ≤ 3 Million/mL or Azoospermia When Using a Daily Regimen of Nestorone® Gel (0, 8 or 12 mg) and Testosterone Gel.
Time Frame: 24 Weeks
Measure: Number; unit: participants
Arm/Group | Testosterone Gel 10 g and Nestorone® 0 mg Per Day | Testosterone Gel 10 g and Nestorone® 8 mg Per Day | Testosterone Gel 10 g Plus Nestorone® Gel 12 mg Per Day
Number analyzed (Participants) | 22 | 18 | 16
participants | 5 | 15 | 14

3. Secondary Outcome: The Number of Men Who Have Azoospermia
Time Frame: 24 Weeks
Measure: Number; unit: participants
Arm/Group | Testosterone Gel 10 g and Nestorone® 0 mg Per Day | Testosterone Gel 10 g and Nestorone® 8 mg Per Day | Testosterone Gel 10 g Plus Nestorone® Gel 12 mg Per Day
Number analyzed (Participants) | 22 | 18 | 16
participants | 5 | 14 | 11

4. Secondary Outcome: The Impact on Sperm Motility in Men Who Are Not Azoospermic Azoospermic.
Time Frame: 24 Weeks
Population: Only subjects with the appropriate amount of data for measurement are represented in the outcome measure data table.
Measure: Mean (Standard Deviation); unit: percentage of sperm
Arm/Group | Testosterone Gel 10 g and Nestorone® 0 mg Per Day | Testosterone Gel 10 g and Nestorone® 8 mg Per Day | Testosterone Gel 10 g Plus Nestorone® Gel 12 mg Per Day
Number analyzed (Participants) | 20 | 7 | 8
percentage of sperm
  Percent Progressive (week 24) | 52.8 (10.70) | 31.9 (26.89) | 29.6 (17.15)
  Percent Non Progressive (week 24) | 10.4 (10.72) | 7.4 (11.94) | 8.3 (4.82)

5. Secondary Outcome: The Impact on Sperm Morphology in Men Who Are Not Azoospermic
Time Frame: 24 weeks
Population: Only subjects with the appropriate amount of data for measurement are represented in the outcome measure data table.
Measure: Mean (Standard Deviation); unit: percentage normal morphology
Arm/Group | Testosterone Gel 10 g and Nestorone® 0 mg Per Day | Testosterone Gel 10 g and Nestorone® 8 mg Per Day | Testosterone Gel 10 g Plus Nestorone® Gel 12 mg Per Day
Number analyzed (Participants) | 21 | 6 | 8
percentage normal morphology | 12.3 (3.87) | 10.8 (4.83) | 9.1 (4.64)

ADVERSE EVENTS:
Arm/Group | Testosterone Gel 10 g and Nestorone® 0 mg Per Day | Testosterone Gel 10 g and Nestorone® 8 mg Per Day | Testosterone Gel 10 g Plus Nestorone® Gel 12 mg Per Day
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/33 | 0/34
Other Adverse Events (participants affected / at risk) | 22/32 | 23/33 | 24/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone Gel 10 g and Nestorone® 0 mg Per Day (N=32) | Testosterone Gel 10 g and Nestorone® 8 mg Per Day (N=33) | Testosterone Gel 10 g Plus Nestorone® Gel 12 mg Per Day (N=34)
Iron Deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Pinguecula (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Stomach Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Application site discolouration (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0
Energy Increased (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 1 | 0
Irritability (General disorders) | 1 | 1 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 2 | 0 | 0
Multiple allergies (Immune system disorders) | 1 | 0 | 0
Seasonal Allergy (Immune system disorders) | 0 | 2 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 1
Genital infection fungal (Infections and infestations) | 0 | 0 | 1
Gonorrhoea (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 3 | 4 | 1
Nasopharyngitis (Infections and infestations) | 7 | 4 | 7
Onychomycosis (Infections and infestations) | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 1
Oropharyngeal gonococcal infection (Infections and infestations) | 0 | 1 | 0
Pareonychia (Infections and infestations) | 0 | 1 | 0
Pharyngitis bacterial (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Tinea versicolour (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 3
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Drug administration error (Injury, poisoning and procedural complications) | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post traumatic pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 1 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 1 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 1
Blood iron decreased (Investigations) | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 1 | 0
Blood triglycerides increased (Investigations) | 1 | 1 | 0
Body temperature fluctuation (Investigations) | 0 | 1 | 0
Heart rate increased (Investigations) | 0 | 0 | 1
semen volume increased (Investigations) | 0 | 0 | 1
Sperm count increased (Investigations) | 0 | 1 | 0
Transaminases increased (Investigations) | 1 | 0 | 0
Weight increased (Investigations) | 1 | 4 | 2
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
headache (Nervous system disorders) | 9 | 6 | 2
Somnolence (Nervous system disorders) | 0 | 1 | 0
aggression (Psychiatric disorders) | 0 | 0 | 1
Anorgasmia (Psychiatric disorders) | 0 | 1 | 0
depressed mood (Psychiatric disorders) | 0 | 1 | 0
depression (Psychiatric disorders) | 1 | 0 | 1
Libido decreased (Psychiatric disorders) | 1 | 2 | 0
insomnia (Psychiatric disorders) | 2 | 2 | 2
libido increased (Psychiatric disorders) | 0 | 0 | 1
mood altered (Psychiatric disorders) | 0 | 1 | 0
mood swings (Psychiatric disorders) | 0 | 2 | 1
nightmare (Psychiatric disorders) | 0 | 1 | 0
dysuria (Renal and urinary disorders) | 0 | 1 | 0
pollakiuria (Renal and urinary disorders) | 0 | 1 | 0
ejaculation disorder (Reproductive system and breast disorders) | 0 | 1 | 0
genital rash (Reproductive system and breast disorders) | 1 | 0 | 0
gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 1
nipple pain (Reproductive system and breast disorders) | 1 | 0 | 0
varicocele (Reproductive system and breast disorders) | 0 | 0 | 1
asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2
postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
acne (Skin and subcutaneous tissue disorders) | 9 | 7 | 5
dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
heat rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
mole excision (Surgical and medical procedures) | 0 | 0 | 1
oral surgery (Surgical and medical procedures) | 1 | 0 | 0
tooth repair (Surgical and medical procedures) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No